CLINICAL TRIAL: NCT00300781
Title: Phase 2 Study of HKI-272 In Subjects With Advanced Breast Cancer
Brief Title: Study Evaluating HKI-272 (Neratinib) In Subjects With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-201 / B1891012
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Breast Neoplasms; Neoplasms
Keywords: phase 2; HER2+ breast cancer; monotherapy neratinib; HKI-272; Neratinib; Nerlynx; PB-272
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neratinib 240 mg, with prior trastuzumab (Experimental): Neratinib administered with 80 mg capsules and 40 mg coated tablets taken orally in prescribed dose of 240 mg daily, as long as tolerated and disease does not worsen.
  Interventions: Drug: neratinib
- Neratinib 240 mg, no prior trastuzumab (Experimental): Neratinib administered with 80 mg capsules and 40 mg coated tablets taken orally in prescribed dose of 240 mg daily, as long as tolerated and disease does not worsen.
  Interventions: Drug: neratinib

INTERVENTIONS:
Drug: neratinib
  Other Names: Nerlynx; HKI-272

SUMMARY:
The purpose of this study is to learn whether neratinib is safe and effective in treating women with advanced human epidermal growth factor receptor 2 (HER2) positive breast cancer.

DETAILED DESCRIPTION:
Arm A: HER2 gene amplification and disease progression following at least 6 weeks of standard doses of Herceptin; Arm B: HER2 gene amplification and no prior Herceptin or HER2-targeted treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of breast cancer and current stage IIIB, IIIC, or IV
* Progression following at least 6 weeks of standard doses of Herceptin (Arm A only)
* Over-expression of HER2
* Tumor tissue available and adequate for analysis at screening
* At least one measurable lesion

Exclusion Criteria:

* Prior treatment with Herceptin (Arm B only)
* More than 4 prior cytotoxic chemotherapy regimens
* Subjects with bone or skin as the only site of measurable disease
* Inadequate cardiac function
* Major surgery, chemotherapy, radiotherapy, investigational agents or other cancer therapy within 1 week of treatment day 1
* Active central nervous system metastases
* Pregnant or breastfeeding women
* Inability to swallow the HKI-272 capsules

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 136 (Actual)
Dates: Start 2006-08-04 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (33):
- United States (13):
  - University of Colorado Hospital, Aurora, Colorado
  - Midwestern Regional Medical Center, Zion, Illinois
  - Louisiana State University, Shreveport, Louisiana
  - The Cancer Center at GBMC, Baltimore, Maryland
  - Oncology Care Associates, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - Norris Cotton Cancer Center Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Virginia Mason Medical Center, Seattle, Washington
- Belgium (3):
  - Institut Jules Bordet Unite du Chimiotherapie, Brussels
  - University Hospital Gasthuisberg, Leuven
  - St-Augustinus Ziekenhuis Oncology Department, Wilrijk
- China (4):
  - The Hospital Affiliated Academy Military Medical Science, Chinese People's Liberation Army, Beijing, Beijing Municipality
  - No. 81 Hospital of Chinese People's Liberation Army, Nanjing, Jiangsu
  - Cancer Hospital Peking Union Medical College, Beijing
  - Chinese People's Liberation Army General Hospital, Beijing
- Institut Gustave ROUSSY Service de Pathologie Mammaire, Villejuif, France
- India (4):
  - Jehangir Clinical Development Centre, Pune, Maharashtra
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra
  - Nizam's Institute of Medical Sciences, Hyderabad, Panjagutta
  - Tata Memorial Centre, Mumbai, Parel
- Mexico (3):
  - Hospital Regional Lic. Adolfo Lopez Mateos Oncología Médica, Mexico City
  - Arke Estudios Clínicos S.A. de C.V., Mexico City
  - Hospital de Especialidades MIG, Mexico City
- Russia (5):
  - N.N. Blokhin Russian Cancer Research Center of RAMS, Moscow
  - Medical Radiological Research Center of RAMS, Department of Radiation and Surgical Methods, Obninsk
  - City Oncology Dispensary, Saint Petersburg
  - City Hospital N 31 Oncology Haematology Dept. For Adults, Saint Petersburg
  - Breast Tumor Department, N.N. Petrov Research Institute of Oncology, Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib 240, Prior Trastuzumab: Neratinib: 80mg capsules and 40mg coated tablets taken orally in prescribed dose of 240mg daily, as long as tolerated and disease does not worsen, in participants with prior trastuzumab treatment.
- Neratinib 240, No Prior Trastuzumab: Neratinib: 80mg capsules and 40mg coated tablets taken orally in prescribed dose of 240mg daily, as long as tolerated and disease does not worsen in participants with with no prior trastuzumab treatment.
Period: Overall Study
Arm/Group | Neratinib 240, Prior Trastuzumab | Neratinib 240, No Prior Trastuzumab
Started | 66 | 70
Completed | 3 | 8
Not Completed | 63 | 62
Not completed — Disease Progression | 55 | 52
Not completed — Adverse Event | 5 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Not Recorded | 0 | 1
Not completed — Symptomatic Deterioration | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated subjects
Groups:
- Neratinib 240, Prior Trastuzumab: Neratinib: 80mg capsules and 40mg coated tablets taken orally in prescribed dose of 240mg daily, as long as tolerated and disease does not worsen in participants with prior trastuzumab treatment.
- Neratinib 240, No Prior Trastuzumab: Neratinib: 80mg capsules and 40mg coated tablets taken orally in prescribed dose of 240mg daily, as long as tolerated and disease does not worsen in participants with no prior trastuzumab treatment.
- Total: Total of all reporting groups
Arm/Group | Neratinib 240, Prior Trastuzumab | Neratinib 240, No Prior Trastuzumab | Total
Number analyzed (Participants) | 66 | 70 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.62 (10.67) | 49.64 (9.92) | 50.60 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 70 | 136
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 52 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 55 | 15 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: 16-week Progression Free Survival
Description: 16 week progression-free survival (PFS) rate of neratinib in women with human epidermal growth factor receptor 2 (HER2) positive breast cancer, either with prior trastuzumab or no prior trastuzumab therapy, evaluated by independent assessment of tumor scans collected at baseline and then every 8 weeks.
Time Frame: From first dose to 16 weeks
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib 240, Prior Trastuzumab | Neratinib 240, No Prior Trastuzumab
Number analyzed (Participants) | 66 | 70
percentage of participants | 58.2 [45.3 to 71.2] | 77.8 [67.6 to 88.1]

2. Secondary Outcome: Objective Response Rate
Description: Percentage of participants with Partial Response (PR) or Complete Response (CR) by independent assessment of tumor per Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From first dose date to progression or last tumor assessment, up to 46 months
Population: Intent to Treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib 240, Prior Trastuzumab | Neratinib 240, No Prior Trastuzumab
Number analyzed (Participants) | 66 | 70
percentage of participants | 24.2 [14.5 to 36.4] | 52.9 [40.6 to 64.9]

3. Secondary Outcome: Clinical Benefit Rate
Description: Percentage of participants who experienced Complete Response (CR), Partial Response (PR), or Stable Disease (SD) ≥ 24 weeks by independent assessment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From first dose date to progression or last tumor assessment, up to 46 months
Population: Intent to Treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib 240, Prior Trastuzumab | Neratinib 240, No Prior Trastuzumab
Number analyzed (Participants) | 66 | 70
percentage of participants | 31.8 [20.9 to 44.4] | 62.9 [50.5 to 74.1]

4. Secondary Outcome: Duration of Response
Description: Number of weeks between Complete Response (CR) or Partial Response (PR) and the first date of disease progression (PD) or death per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: From start date of response to first PD/death, up to 46 months
Population: Subjects in Intent to Treat population with CR or PR
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Neratinib 240, Prior Trastuzumab | Neratinib 240, No Prior Trastuzumab
Number analyzed (Participants) | 16 | 37
weeks | 40.3 [32.3 to 80.1] | 60.0 [40.1 to 100.1]

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose, up to 46 months.
Arm/Group | Neratinib 240, Prior Trastuzumab | Neratinib 240, No Prior Trastuzumab
Serious Adverse Events (participants affected / at risk) | 19/66 | 17/70
Other Adverse Events (participants affected / at risk) | 66/66 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 240, Prior Trastuzumab (N=66) | Neratinib 240, No Prior Trastuzumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 6
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 240, Prior Trastuzumab (N=66) | Neratinib 240, No Prior Trastuzumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 4 | 8
Leukopenia (Blood and lymphatic system disorders) | 4 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 19 | 6
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 63 | 64
Dry mouth (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 7
Haemorrhoids (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 27 | 23
Stomatitis (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 16 | 23
Asthenia (General disorders) | 3 | 10
Fatigue (General disorders) | 26 | 7
Oedema peripheral (General disorders) | 4 | 5
Pyrexia (General disorders) | 5 | 12
Nasopharyngitis (Infections and infestations) | 2 | 5
Paronychia (Infections and infestations) | 0 | 6
Urinary tract infection (Infections and infestations) | 7 | 1
Alanine aminotransferase increased (Investigations) | 1 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 5
Weight decreased (Investigations) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 15 | 12
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7
Dizziness (Nervous system disorders) | 5 | 6
Dysgeusia (Nervous system disorders) | 6 | 0
Headache (Nervous system disorders) | 12 | 14
Insomnia (Psychiatric disorders) | 3 | 4
Dysuria (Renal and urinary disorders) | 1 | 6
Pollakiuria (Renal and urinary disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 4
Rash (Skin and subcutaneous tissue disorders) | 14 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less